CLINICAL TRIAL: NCT01762605
Title: Supportive Care Versus Casting for Distal Forearm Buckle Fractures in Children; A Randomized Controlled Trial
Brief Title: Treatment of Distal Radius Buckle Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inadequate enrollment
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00012567
Record Dates: First submitted 2013-01-03; First posted 2013-01-08 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2018-08

CONDITIONS: Fracture Treatment
MeSH Terms: interventions — Palliative Care; POLR1G protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive Care (Experimental): No casting or splinting, supportive care only by parents
  Interventions: Other: Supportive Care
- Cast (Active Comparator): Casting for 4 weeks
  Interventions: Procedure: Cast

INTERVENTIONS:
Other: Supportive Care
  Arms: Supportive Care
Procedure: Cast
  Arms: Cast

SUMMARY:
This study determines if patients with buckle fractures of the distal radius and/or ulna treated with supportive care only demonstrate non-inferior outcomes in regard to pain control during healing, functional outcome at the wrist joint, and parental satisfaction, when compared with patients treated with the standard treatment regimen of 3-4 weeks in a short arm cast.

ELIGIBILITY:
Inclusion Criteria:

Children age 1-17 with buckle fractures of the distal radius and/or ulna. -

Exclusion Criteria:

* Patients are excluded if there is any other injury to the upper limb or serious bodily trauma that might complicate pain scores. Children with suspected or proven metabolic bone disease, or pathologic fractures are excluded due to resultant abnormal bone healing.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pain | 4-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Frino, MD, Principal Investigator — Atrium Health Wake Forest Baptist